CLINICAL TRIAL: NCT02398851
Title: TacTIC- Trans-disciplinary Chronic Disease Continuity of Care Model
Acronym: TacTIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro 5429
Record Dates: First submitted 2015-03-06; First posted 2015-03-26 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Chronic Disease; Geriatrics
MeSH Terms: conditions — Chronic Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TacTIC care model (Other): Compare the 30-day readmission rate in adult patients who receive care in a trans-disciplinary chronic disease continuity of care model with integrated technology (mobile devices such as tablets, iPads and smartphones)
  Interventions: Behavioral: TacTic care model
- Standard of Care (Other): Compare standard practice (patient-centered, coordinated care model without the integration of technology
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: TacTic care model — Patients receive care in a trans-disciplinary chronic disease continuity of care model integrated with technology (mobile devices such as tablets, iPads and smartphones
  Arms: TacTIC care model
Behavioral: Standard of care — Patients receive care in a patient-centered, coordinated care model without the integration of technology
  Arms: Standard of Care

SUMMARY:
The overall aim of this study is to create a trans-disciplinary chronic disease continuity of care model with health information technology, utilizing mobile devices such as tablets, iPads and smartphones.

DETAILED DESCRIPTION:
This study aims to explore if a trans-disciplinary chronic disease continuity of care model with integrated technology (mobile devices such as tablets, iPads and smartphones) to standard practice (patient-centered, coordinated care model without the integration of technology) will results in a reduction in 30-day readmission rate in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients on a 43 bed medical surgical unit
* Adult patients on 44 bed geriatric unit

Exclusion Criteria:

* Adult patients admitted and not diagnosed with chronic disease
* Patients who are transferred between Intervention and non-Intervention unit
* Patients who refuse
* Patients with delirium, dementia and altered mental status
* Patients who cannot read and write in any language
* Patients in the intervention group who cannot use mobile technology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Reduction in the 30-day readmission rates in adult patients who receive care in a trans-disciplinary chronic disease continuity of care model integrated with technology (mobile devices such as tablets, iPads and smartphones). | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Julius Gardin, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical center, Hackensack, New Jersey, United States